CLINICAL TRIAL: NCT03337581
Title: The Safety、Efficacy and Pharmacokinetics of Dexmedetomidine Administered Through Different Routes in Pediatric
Brief Title: Pharmacodynamics and Pharmacokinetics of Dexmedetomidine in Pediatric
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Medical Association (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: No.2017-62
Record Dates: First submitted 2017-09-01; First posted 2017-11-09 (Actual); Last update posted 2017-11-09 (Actual); Status verified 2017-08

CONDITIONS: Pediatrics; Dexmedetomidine; Pharmacodynamics; Pharmacokinetics
Keywords: Dexmedetomidine; pediatrics; Pharmacodynamics; Pharmacokinetics
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- group 1.1 (Sham Comparator): Normal saline group
  Interventions: Drug: Dexmedetomidine
- group 1.2 (Experimental): 0.25μg/kg dexmedetomidine group
  Interventions: Drug: Dexmedetomidine
- group 1.3 (Experimental): 0.5μg/kg dexmedetomidine group
  Interventions: Drug: Dexmedetomidine
- group 1.4 (Experimental): 0.75μg/kg dexmedetomidine group
  Interventions: Drug: Dexmedetomidine
- group 1.5 (Experimental): 1.0μg/kg dexmedetomidine group
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — see arms

SUMMARY:
1. Acute Hemodynamic and respiratory Changes After Rapid Intravenous different doses of Dexmedetomidine in Pediatric.
2. Pharmacokinetics after a single Rapid Intravenous dose of Dexmedetomidine in Pediatric.
3. Pharmacokinetics after a single dose of Dexmedetomidine administered as a nasal spray in Pediatric.

ELIGIBILITY:
Inclusion Criteria:

* selective operation of inguinal hernia repair、orthopedics operation or general surgery operation in children
* aged 3-9 years
* ASA I - II
* enter the operating room by himself without parents
* normal liver and kidney function
* no history of anesthesia medication allergy.

Exclusion Criteria:

* allergic to dexmedetomidine, similar active ingredients or excipients
* G-6-PD deficiency
* a history of arrhythmia, bronchial and cardiovascular diseases, abnormal liver function and so on
* a history of use of alpha 2 receptor agonists or antagonists.

Ages: 3 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 187 (Estimated)
Dates: Start 2017-10-20 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Acute Hemodynamic and respiratory Changes After Rapid Intravenous of Dexmedetomidine | up to 4 months
  Acute Hemodynamic and respiratory Changes After Rapid Intravenous different doses of Dexmedetomidine in Pediatric
Pharmacokinetics after a single Rapid Intravenous dose of Dexmedetomidine in Pediatric | up to 6 months
  After a single Rapid Intravenous dose of Dexmedetomidine in Pediatric，blood samples will be collected ,and dexmedetomidine plasma concentrations were measured with High Performance Liquid Chromatography-Tandem Mass Spectrometry (HPLC-MS/MS).
Pharmacokinetics of Dexmedetomidine administered as a nasal spray | up to 6 months
  After a single dose of Dexmedetomidine administered as a nasal spray in Pediatric,blood samples will be collected ,and dexmedetomidine plasma concentrations were measured with High Performance Liquid Chromatography-Tandem Mass Spectrometry (HPLC-MS/MS).

CONTACTS AND LOCATIONS:
Overall Officials: Huacheng Liu, Study Director — The Second Affiliated Hospital and Yuying Children's Hospital of Wenzhou Medical University
Locations (1):
- The second Affiliated Hospital and Yuying Children's Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China

DOCUMENTS (3):
  • Study Protocol (2017-10-12): https://cdn.clinicaltrials.gov/large-docs/81/NCT03337581/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-12): https://cdn.clinicaltrials.gov/large-docs/81/NCT03337581/SAP_001.pdf
  • Informed Consent Form (2017-10-12): https://cdn.clinicaltrials.gov/large-docs/81/NCT03337581/ICF_002.pdf